CLINICAL TRIAL: NCT06484218
Title: Guided Endodontics Compared to Conventional Endodontic Treatment in Calcified Lower Incisors: a Comparative in Vivo Pilot Study.
Brief Title: Guided Endodontics Compared to Conventional Endodontic Treatment in Calcified Lower Incisors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USJ-2023-214
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Dentinal Loss
Keywords: Lower incisors; pulp canal calcification; guided endodontics; dentinal loss; treatment duration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CET (Experimental): The CET presented the conventional endodontic technique where one incisor was treated under microscope with an ultrasonic tip.
  Interventions: Procedure: conventional endodontic treatment; Procedure: Guided endodontic treatment
- Group GET (Active Comparator): The GET presented the guided endodontic technique where one incisor was treated with a surgical guide.
  Interventions: Procedure: conventional endodontic treatment; Procedure: Guided endodontic treatment

INTERVENTIONS:
Procedure: conventional endodontic treatment — The conventional access cavity was prepared under the microscope through the incisal edge as this approach facilitates straight-line access. A high-speed contra-angle handpiece, associated with a long surgical bur 010 (Meisinger, CO, USA), was used until the dentin was exposed, which is in general 3 to 4 millimeters from the incisal edge. Then, the ultrasonic tip ED5 (woodpecker-DTE, Guilin, China) was marked with a stopper according to the calcification level viewed on the preoperative CBCT and then used gently at the stopper level until the canal was found.
Procedure: Guided endodontic treatment — In all cases, digital and clinical protocols were followed according to the method reported by Zehnder et al. and Connert et al. The guide was replaced, and the access cavity precisely drilled using the EG6 drill, mounted on a low-speed contra-angle handpiece. With every 3 mm of progression, the cavity was rinsed, and the head of the bur was cleaned until reaching the canal. The irrigation was done to avoid overheating the dentine and the accumulation of dentine debris

SUMMARY:
The dental pulp is a vital tissue that can be prone to physiological or pathological changes. Denticles, pulp stones, or other calcifications are frequently observed within "healthy" pulps. However, these tissue alterations can complicate the endodontic treatment. According to the American Association of Endodontists, teeth exhibiting "pulpal obliteration" fall into the moderate to high difficulty category of treatments, and their failure rate ranges from 10 to 19 per cent 1,2. In fact, pulpal calcification alone is not a reason for endodontic treatment. Root canal treatment is recommended and deemed necessary only in the presence of peri-radicular pathology or if the affected tooth shows symptoms. Today's techniques and materials offer higher standards, resulting in better root canal treatments and allowing proper handling of procedural errors. One of these materials is Cone beam computed tomography (CBCT) which is more reliable in detecting periapical lesions compared with digital periapical radiographs 3,visual aids, and ultrasonics 1. However, when performed by a non-experienced dentist, the risk of perforations, missed canals, stripping, and ledges arises 2. For the treatment of these challenging instances, the development of guided endodontics with a trephination guide, a metal sleeve, and an appropriate drill might be of interest 4. With several in vitro studies 5-7 and case reports 8,9 being published each year, this approach is becoming more prevalent in the literature. Additionally, a new endodontic guide software is being used to build new shapes for guides, sleeves, and drills, which will make it easier to attain correct access using the guiding technique. However, there is no information regarding the detection and negotiation of root canals, the dental substance loss, the treatment duration using the guided technique compared to the conventional technique for root canal treatments (RCTs) in clinical practice 10. This study is conducted to compare the conventional endodontic treatment to the guided approach in lower incisors with calcified root canals by focusing on the following aspects: the detection and negotiation of canals, the amount of substance loss, and the treatment duration.

DETAILED DESCRIPTION:
Seven patients having two calcified lower incisors requiring root canal treatment were selected. For each patient, one incisor was treated with the CET while the other incisor was treated with the GET by a single operator, a graduate endodontic resident. The intracanal space of the treated teeth was volumetrically measured and compared using the indirect post core technique and Blenderfordental software (version 3.3 lts). The time was recorded from the start of the treatment until the root canal was negotiated to determine the treatment duration. Various statistical tests including BM SPSS Statistics software version 25.0 and the Wilcoxon signed rank test were used to identify potential significant differences between the CET and the GET in terms of volume and treatment duration with a significance threshold set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Single-rooted mandibular incisor.
2. Pulp canal obliteration extended from the cementoenamel junction more than five millimeters to the radicular pulp canal space.
3. Vertucci type 1 classification.
4. Teeth needing endodontic intervention: symptomatic tooth, peri-radicular lesion or endodontic-periodontic lesion.
5. Straight root canal: curvature less than five degrees.
6. No mobility.

Exclusion Criteria:

1. Mandibular incisor with two roots.
2. Teeth treated with a crown.
3. Severely carious teeth.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Amount of dental substance loss | 24 hours
  Regarding the substance loss, the CET resulted in higher intracanal volume compared to the GET (7.8±3.3 mm3 vs 5.3±1.3 mm3, p=0.018).
the detection and negotiation of canals | 24 hours
  Seven teeth were treated using the CET (n=7) and another seven using the GET (n=7). All teeth had negotiable canals except for one which was treated using the CET having the calcification level at the third third level of the middle part. . This unsuccessful case was referred to microsurgery treatment.
the treatment duration | 24 hours
  the CET presented a significantly higher TD compared to the GET (69.0±57.4 mins vs 14.1±8.2 mins; p=0.018).

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No